CLINICAL TRIAL: NCT01050400
Title: CYP2D6 Screening for Adverse Drug Reactions to Codeine in Breast Milk
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: R-09-442
Record Dates: First submitted 2010-01-11; First posted 2010-01-15 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Cytochrome P450 2D6 Ultra-rapid Metabolism
Keywords: CYP2D6; Genetic Polymorphism; codeine; breastfeeding
MeSH Terms: conditions — Breast Feeding | interventions — Cytochrome P-450 CYP2D6; Genetic Testing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva and breast milk samples.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Observant: Individuals within this group will receive pharmacotherapy according to the established institutional guidelines.
  Interventions: Genetic: Cytochrome P450 2D6 (CYP2D6) genetic screening.
- Prospective CYP2D6 genetic screening: Individuals within the prospective group will receive their CYP2D6 genotype results prior to pharmacotherapy and their analgesic regimen will be tailored to their genetic results.
  Interventions: Genetic: Cytochrome P450 2D6 (CYP2D6) genetic screening.

INTERVENTIONS:
Genetic: Cytochrome P450 2D6 (CYP2D6) genetic screening. — Genetic screening for cytochrome P450 2D6 (CYP2D6) polymorphism will be conducted on genetic information obtained from non-invasive salivary samples.

SUMMARY:
The purpose of this study is to determine if non-invasive salivary genetic screening of breastfeeding mothers taking codeine will allow for the successful identification of mother-infant pairs susceptible to adverse events and to prevent these adverse events by personalizing their medication to their genetics.

DETAILED DESCRIPTION:
Currently, the opioid analgesic codeine is commonly administered to breastfeeding mothers after Caesarean section for pain relief. Codeine was originally considered safe to use while breastfeeding however, increased risk of adverse drug reactions has been demonstrated in mothers taking codeine, as well as their breastfed infants, when the mother possesses a genetic variation resulting in cytochrome P450 2D6 (CYP2D6) ultra-rapid metabolizer (UM) phenotype. On average, most people convert about 10-15% of their codeine dose to morphine resulting in pain relief however, UM individuals can convert up to 50% of their codeine doses into active morphine. As many as 4% of North Americans may be UMs and these mothers and their breastfed infants are at high risk of serious adverse events despite "safe" codeine dosing due to morphine overproduction and accumulation in the mother and her breast milk. Observed side effects include severe sedation, decreased rate and depth of breathing and even infant death. In response to this problem, our hospital-based clinical trial strives to identify at-risk UM mother-infant pairs by performing a genetic test on non-invasive, voluntary saliva samples from mothers giving birth by Caesarean section and who will need codeine for pain relief while breastfeeding. We believe that this test will allow us to reliably identify at-risk UM mother-infant pairs and prevent adverse drug reactions in both by tailoring analgesic therapy to their genetic results: mothers identified as being UMs will be given other suitable analgesics, such as ibuprofen, in place of codeine-containing preparations. We propose that this prospective study will generate high-level data supporting the cost-effective genetic screening of mothers who will be taking codeine while breastfeeding before they begin taking their medications. Such testing is currently possible on a nation-wide scale through collaboration with the Canadian Pharmacogenomics Network for Drug Safety (CPNDS).

ELIGIBILITY:
Inclusion Criteria:

Women who:

* Have a pre-scheduled Caesarean section
* Provide DNA for CYP2D6 genetic analysis
* Breastfeed their infants
* Take codeine-containing medication during breastfeeding (retrospective screening group and non-CYP2D6 ultrarapid metabolizers in prospective screening group)

Exclusion Criteria:

* Mothers who do not provide consent prior to Caesarian section surgery
* Mothers who take other sedative medications besides codeine during breastfeeding (these include benzodiazepines, skeletal muscle relaxants, psychotropic agents).

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women undergoing elective caesarian section surgery and planning to breastfeed while concurrently taking codeine for post-partum pain relief within St. Joseph's Hospital in London and St. Michael's Hospital in Toronto.
Sampling Method: Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2009-02-24 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2012-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of maternal and neonatal CNS depression in the prospective pharmacogenetic screening group to that of a retrospectively screened population | 5-8 days post c-section surgery

SECONDARY OUTCOMES:
Incidence of the phase II uridine diphosphate glucuronyltransferase 2B7 (UGT2B7)*2/*2 variant which has been associated with higher morphine 6-glucuronide to morphine ratios. | Minimum 1 week prior to c-section
Incidence of the C3435T polymorphism in the multi-drug resistance gene (MDR1) which has been associated with significantly greater pain relief from morphine treatment. | Minimum 1 week prior to c-section
Incidence of the A118G polymorphism in the opioid receptor 1 (OPRM1) which has been associated with reduced response to morphine treatment. | Minimum 1 week prior to c-section

CONTACTS AND LOCATIONS:
Overall Officials: Gideon Koren, MD, Principal Investigator — Western University, Canada
Locations (1):
- St. Joseph's Hospital, London, Ontario, Canada